CLINICAL TRIAL: NCT01405547
Title: Impact of Maternal Metabolic Abnormalities in Pregnancy on Human Milk and Subsequent Infant Metabolic Development
Brief Title: Gestational Metabolic Abnormalities and Maternal and Infant Nutrition and Health
Status: Completed | Type: Observational
Sponsor: Anthony Hanley (Other)
Collaborators: Canadian Diabetes Association (Other); Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Sponsor-Investigator, Anthony Hanley, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: 488057
Record Dates: First submitted 2011-07-12; First posted 2011-07-29 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes; Hyperglycemia; Insulin Resistance; Obesity
Keywords: Gestational Diabetes; Gestational Hyperglycemia; Gestational Insulinemia; Maternal Obesity; Human Milk; Lactogenesis; Obstetrics; Nutrition; Infant Growth
MeSH Terms: conditions — Diabetes, Gestational; Hyperglycemia; Insulin Resistance; Obesity; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Childhood obesity is on the rise and is a major risk factor for type 2 diabetes later in life. Recent evidence indicates that abnormalities that increase risk for diabetes may be initiated early in infancy. Since the offspring of women with diabetes have an increased long-term risk for obesity and type 2 diabetes, the impact of maternal metabolic abnormalities on early nutrition and infant metabolic trajectories is of considerable interest. The purpose of the study is to investigate the impact of maternal nutrition and metabolic abnormalities in pregnancy on human milk and subsequently on infant health over the first year of life.

DETAILED DESCRIPTION:
The current investigation is a prospective study conducted within ongoing cohort studies of women and their offspring. Pregnant women attending outpatient obstetrics clinics in Toronto, Canada are recruited. The overall study protocol includes four study visits between the second half of pregnancy and the first year of infant's life and interim phone call interviews:

* Pregnant women undergo an oral glucose tolerance test at an expected average of 30 weeks of gestation and complete medical and lifestyle questionnaires including food frequency questionnaires.
* Infant birth anthropometry measurements and human milk samples are collected at an expected average of 3 days postpartum. The timing of onset of lactogenesis II is asked at 3d, 5d, 7d postpartum or until the event occurrence up to day 7.
* At 3 months postpartum, follow-up assessments including infant anthropometry, medical and lifestyle questionnaires and human milk sample collection are completed.
* Interim telephone interviews are conducted at 6 weeks and 5, 7, 9 months postpartum to characterize infant feeding and supplementation behaviors.
* At 12 months postpartum, infant anthropometric assessments are conducted.

ELIGIBILITY:
Inclusion Criteria:

* singleton or twin pregnancy
* aged 20 years or older at the time of recruitment
* intention to breastfeed

Exclusion Criteria:

* pre-existing diabetes

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women are recruited in outpatient clinic waiting areas at Mount Sinai Hospital in Toronto, Canada, a large tertiary care centre.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Infant growth | Growth from birth to anthrometry at 12mo

SECONDARY OUTCOMES:
Human milk composition | At 3d and at 3mo postpartum
Onset of lactogenesis II | At 3d, 5d, 7d postpartum until the event occurrence of milk-coming-in up to day 7.
  If the participant reports no milk-coming-in at the day 7 postpartum interview, the response is recorded as no milk-coming-in by day 7 postpartum.
Gestational diabetes | An expected average of 30 weeks of gestation
Gestational metabolic abnormalities | An expected average of 30 weeks of gestation
Getational hyperglycemia and insulinemia (insulin resistance/sensitivity) | An expected average of 30 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hanley, PhD, Study Chair — University of Toronto; Sylvia Ley, PhD, Study Director — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ley SH, O'Connor DL, Retnakaran R, Hamilton JK, Sermer M, Zinman B, Hanley AJ. Impact of maternal metabolic abnormalities in pregnancy on human milk and subsequent infant metabolic development: methodology and design. BMC Public Health. 2010 Oct 6;10:590. doi: 10.1186/1471-2458-10-590. PMID 20925937
- [Result] Ley SH, Hanley AJ, Sermer M, Zinman B, O'Connor DL. Associations of prenatal metabolic abnormalities with insulin and adiponectin concentrations in human milk. Am J Clin Nutr. 2012 Apr;95(4):867-74. doi: 10.3945/ajcn.111.028431. Epub 2012 Feb 29. PMID 22378730
- [Result] Ley SH, Hanley AJ, Retnakaran R, Sermer M, Zinman B, O'Connor DL. Effect of macronutrient intake during the second trimester on glucose metabolism later in pregnancy. Am J Clin Nutr. 2011 Nov;94(5):1232-40. doi: 10.3945/ajcn.111.018861. Epub 2011 Sep 28. PMID 21955650
- [Derived] LeMay-Nedjelski L, Butcher J, Ley SH, Asbury MR, Hanley AJ, Kiss A, Unger S, Copeland JK, Wang PW, Zinman B, Stintzi A, O'Connor DL. Examining the relationship between maternal body size, gestational glucose tolerance status, mode of delivery and ethnicity on human milk microbiota at three months post-partum. BMC Microbiol. 2020 Jul 20;20(1):219. doi: 10.1186/s12866-020-01901-9. PMID 32689933
- [Derived] Ley SH, Hanley AJ, Sermer M, Zinman B, O'Connor DL. Lower dietary vitamin E intake during the second trimester is associated with insulin resistance and hyperglycemia later in pregnancy. Eur J Clin Nutr. 2013 Nov;67(11):1154-6. doi: 10.1038/ejcn.2013.185. Epub 2013 Sep 25. PMID 24065066